CLINICAL TRIAL: NCT05878652
Title: Utilization of a 3D Printed Customized Knee Extender on Patient Outcomes Following ACL Injuries
Brief Title: Playmaker 3D Printed Knee Extender
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study structure was flawed and as a result the investigator had closed the study.
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Playmaker
Record Dates: First submitted 2023-03-28; First posted 2023-05-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: ACL; ACL Injury
Keywords: Desktop 3D Printing; Knee Extender; Pre-habilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants will utilize a 3D printed knee extension device and an at-home prehabilitation program designed to be used with the 3D printed knee extension device.
  Interventions: Device: 3D printed knee extender device
- Control Arm (Other): Participants will receive the standard prehabilitation education at Sanford and provided exercises to do at home.
  Interventions: Other: Standard Prehabilitation Education

INTERVENTIONS:
Device: 3D printed knee extender device — Participants will receive the standard of prehabilitation education at Sanford as well as a 3D printed knee extension device with sealed water bottles and a home prehabilitation program designed to be used with the 3D printed knee extension device.
  Arms: Experimental Arm
Other: Standard Prehabilitation Education — Participants in the control group will receive the standard prehabilitation education at Sanford and provided exercises to do at home.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to explore the development of, and patient outcomes associated with, the use of individually printed knee extender in conjunction with a video-based home pre-habilitation program for patients who have suffered an ACL rupture before surgery.

DETAILED DESCRIPTION:
The proposed study will assess the efficacy of utilizing desktop 3DP for patient-specific knee extenders paired with a video-based home pre-habilitation program to address the aforementioned barriers. If the novel device and home program is found to be a viable treatment option, this may improve or replace current treatments for knee pre-habilitation, increase accessibility to proper treatment, and reduce cost and time burden on patients, PTs, and providers. The study will offer a greater understanding of potential improvements to clinical workflows and efficiencies through using 3DP. This technology is an under- utilized resource; further research into the applications of 3DP in the field of orthopaedics will provide opportunities to improve patient care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 14-60 years old patients who have suffered an isolated primary ACL rupture

Exclusion Criteria:

* Patients who have already attained full knee extension
* Open skin wounds that would come into contact with the device
* Pregnant women

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Knee Extension Range of Motion | Change from baseline range of motion to day of ACL reconstruction.
  Knee extension range of motion is measured by a trained study member who is blinded to the participant's study group using a goniometer in clinic. Participants are seated on the exam table with their leg maximally extended. The center of the goniometer is placed over the lateral epicondyle of the affected knee. One of the goniometer arms is aimed proximally, pointing toward the greater trochanter of the hip. The other arm is aimed distally, pointing toward the lateral malleolus of the ankle. The study member then reads the angle created by the arms of the goniometer in this position.
Time to Achieve Full Knee Extension | Through study completion, an average of 4 weeks.
  Full knee extension will be measured at home by participants by placing a clicking device under their knee which will produce an audible "click" when the knee is fully extended, and the clicker is depressed. Participants in the control and experimental groups record whether they are able to depress the clicker in at-home logs daily paper logs and online surveys in RedCap, respectively.

SECONDARY OUTCOMES:
Knee Swelling | Through study completion, an average of 4 weeks.
  Participant knee swelling is measured by a trained study member who is blinded to the participant's study group in clinic. Circumference of the knee is used as a proxy for knee swelling, and is measured by wrapping a tape measure around the circumference of the knee just proximal to the superior pole of the patella with resting tension.
Average Daily Pain Level | From baseline until their ACL reconstruction, assessed up to an average of 4 weeks.
  Participant average pain level for control and experimental groups is recorded in an at-home daily paper log and online surveys in RedCap, respectively.
Water Bottles Used with Knee Sling | From baseline until their ACL reconstruction, assessed up to an average of 4 weeks.
  Participants in the experimental group record how many water bottles they use to weigh down their knee sling, up to a maximum of ten water bottles, in online surveys in RedCap in each of the morning, afternoon, and evening prehab sessions.
Minutes Spent Using Knee Sling | Through study completion, an average of 4 weeks.
  Participants in the experimental group record how many minutes they spend using the knee sling, up to a maximum of ten minutes, in online surveys in RedCap in each of the morning, afternoon, and evening prehab sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Skelley, MD, Principal Investigator — Sanford Health
Locations (2):
- United States (2):
  - Sanford Orthopedics and Sports Medicine, Fargo, North Dakota
  - Sanford Orthopedics and Sports Medicine, Sioux Falls, South Dakota